CLINICAL TRIAL: NCT06305962
Title: Phase 0/1 Study of the Safety and Tolerability of 177Lu-RAD204, a Lutetium-177 Radiolabelled Single Domain Antibody Against Programmed Cell Death-Ligand 1 in Patients With Metastatic Solid Tumours
Brief Title: 177Lu-anti-PD-L1 sdAb in Metastatic Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-RAD204.2023.0001
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: PDL1 Gene Mutation; Non Small Cell Lung Cancer; Small Cell Lung Cancer ( SCLC ); TNBC, Triple Negative Breast Cancer; Cutaneous Melanoma; HNSCC; Endometrial Cancer; Mmr Deficiency; MSI-High
Keywords: PDL1 Positive; Non Small Cell Lung Cancer; Small Cell Lung Cancer (SCLC); TNBC, Triple Negative Breast Cancer; Cutaneous Melanoma; HNSCC; Endometrial cancer; Mmr Deficiency; MSI-High
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Melanoma; Squamous Cell Carcinoma of Head and Neck; Endometrial Neoplasms; Turcot syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 177Lu-RAD204 (Experimental): Single-arm, open-label study of 177Lu-RAD204 consisting of a Phase 0 Imaging Period (Im) and a Phase 1 Treatment Period (Tr).
  Interventions: Drug: 177Lu-RAD204

INTERVENTIONS:
Drug: 177Lu-RAD204 — 177Lu-RAD204 administered at Imaging (im) and Treatment (tr) doses

SUMMARY:
This is a Phase 0/1, First-in-Human (FIH), study to evaluate safety, tolerability, biodistribution, radiation dosimetry and preliminary anti-tumour activities of 177Lu-RAD204 in participants with selected solid tumours, to identify the MTDs/ recommended doses of 177Lu-RAD204 for future exploration.

The study will consist of a Pre-screening Period (if applicable for PD-L1 testing), a Screening Period of up to 4 weeks, followed by a Phase 0 (Imaging) Period for imaging and dosimetry to 177Lu-RAD204im and a Phase I (Treatment) Period for 177Lu-RAD204tr dose escalation.

DETAILED DESCRIPTION:
This is a first in human, Phase 0/1, open-label study of 177Lu-RAD204 consisting of an Imaging Period with 177Lu-RAD204im (imaging dose) and a Treatment Period with 177Lu-RAD204tr (treatment dose) to determine the recommended dose(s) for future exploration of 177Lu-RAD204 in participants with PDL1+ advanced solid tumors.

Screening Period: Screening Period of up to 4 weeks. Phase 0 (Imaging Period): Low dose (10mCi) of 177Lu-RAD204 administered on Imaging Day 1 with a follow-up period of up to 2 weeks to assess imaging, safety and dosimetry. The dose may be increased, if needed, to improve image quality.

Phase 1 (treatment Period): 177Lu-RAD204tr dose escalation

* Treatment Period with each cycle lasting 6 weeks. Extension of the planned dose intervals are possible following discussion and agreement between the Sponsor and Investigator.
* Participants may be treated with multiple cycles, as long as they appear to derive clinical benefit as determined by the Investigator and provided there is adequate clinical safety and organ dosimetry data.
* Dose Limiting Toxicity (DLT) observation period for 177Lu-RAD204tr is 6 weeks following the first injection of 177Lu-RAD204tr.
* Should an alternative treatment schedule be explored, the DLT observation period for 177Lu-RAD204tr at that dose level will be the proposed cycle duration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent prior to start of any study procedures and assessments and must be willing to comply with all study procedures.
2. Adult participants ≥ 18 years of age.
3. Participants with a documented history of histopathologically confirmed relapsed/refractory locally advanced, inoperable or metastatic NSCLC, SCLC, TNBC, cutaneous melanoma, HNSCC, endometrial cancer or any cancer that is known to be MMR deficient or MSI high with documented disease progression during or after their most recent line of anticancer therapy. Participants must be refractory to or have refused standard of care therapy (including PD-1/PD-L1 inhibitors) or have refused or have no standard of care therapy available that is likely to provide clinical benefit.
4. Participants with PD-L1 positive NSCLC, SCLC, TNBC, cutaneous melanoma, HNSCC, endometrial cancer or any cancer that is known to be MMR deficient or MSI high:

   * If the participant tumour's PD-L1 expression status is unknown, PD-L1 positivity may be determined in a pre-screening step whereby the participant may be approached to provide written informed consent to have their tumour tissue undergo IHC testing as determined by a validated test (tumour tissue may be obtained from archived samples or from a freshly obtained biopsy).
   * Any number of prior treatment lines are allowed.
5. Must have at least 1 measurable target lesion according to RECIST version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Participants must have a life expectancy of ≥ 4 months in the opinion of the Investigator.
8. Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin (β-hCG) test and must not be breastfeeding. WOCBP are defined as those who are not surgically sterile or post-menopausal. Female participants will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. Female participants < 50 years old who meet the criteria for post-menopausal status without previous surgical sterilisation should be considered for further investigation with luteinising hormone (LH) and follicle stimulating hormone (FSH) levels to confirm serological post-menopausal status.
9. WOCBP must agree to use a highly effective method of contraception during the study and for 14 days after the last injection of 177Lu-RAD204im and/or 6 months after the last dose of 177Lu-RAD204tr, whichever occurs later. Acceptable methods of contraception are described in Section 13.3 of the Protocol.
10. Male participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during the study and for 14 days after the last injection of 177Lu-RAD204im and/or 6 months after the last dose of 177Lu-RAD204tr, whichever occurs later. All male participants must agree to not donate sperm during the study and for 14 days after the last injection of 177Lu-RAD204im and/or 6 months after the last dose of Lu-RAD204tr, whichever occurs later. Acceptable methods of contraception are described in Section 13.3 of the Protocol.
11. Participants with previously treated brain metastases are eligible to participate if:

    * they are neurologically and radiologically stable (no evidence of progression by imaging; same imaging modality [magnetic resonance imaging (MRI) or computed tomography (CT) scan] must be used for each assessment) for at least 28 days prior to the first dose of 177Lu-RAD204im,
    * do not require steroids to treat associated neurological symptoms, and
    * have no history of leptomeningeal disease or spinal cord compression.
    * Participants with active brain metastases who have not received brain-directed therapy such as radiotherapy are not eligible to enroll.
12. For Phase I:

    * Participants must have positive lesion(s) by 177Lu-RAD204im SPECT/CT per central review as described in Image Review Charter, and
    * Participants without any positive lesion by 177Lu-RAD204im SPECT/CT, e.g. due to poor image quality, may be allowed to enrol on a case-by-case basis at the discretion of the Principal Investigator and in discussion with study Sponsor, provided the participant's tumour is known to express PD-L1.

Exclusion Criteria:

1. History of prior organ transplant.
2. Any other known, active malignancy, except for treated cervical intraepithelial neoplasia or non-melanoma skin cancer. Patients with a history of malignancies of low recurrence potential who have received curative-intent therapy may be approved on a case-by-case basis in discussion with study Sponsor, if it is determined not to put the patient at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
3. Have any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures such as participants with severe claustrophobia who are unresponsive to oral anxiolytics, participants with low back pain who cannot lie comfortably on an imaging table, participants who are hyperactive or hyperkinetic such that they cannot tolerate lying still for multiple time point imaging procedures, etc.
4. Residual toxicity ≥ Grade 2 from prior anti-cancer therapy (except alopecia).
5. History of uncontrolled allergic reactions and/or known or expected hypersensitivity to protein therapeutics, 177Lu-RAD204 or any of its excipients.
6. Inadequate organ functions as reflected in laboratory parameters:

   * Creatinine clearance or body surface area (BSA) adjusted estimated glomerular filtration rate (eGFR) (calculated using any clinically validated formula, preferably Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), or measured) < 60 mL/min
   * Platelet count of < 80 × 109/L
   * Absolute neutrophil count (ANC) < 1.5 × 109/L
   * Haemoglobin < 9 g/dL
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × ULN, or > 5 × ULN for patients with known liver metastases
   * Total bilirubin > 1.5 × ULN, except for patients with documented Gilbert's syndrome who are eligible if total bilirubin ≤ 3 × ULN
   * For participants not taking warfarin or other anticoagulants: international normalized ratio (INR) ≥ 1.5 or prothrombin time (PT) ≥ 1.5 × ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≥1.5 × ULN. Participants taking warfarin must be on a stable dose that results in a stable INR < 3.5. Among participants receiving other anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
7. Patients requiring blood product transfusion within 4 weeks of first dose of 177Lu-RAD204tr are not eligible to participate.
8. Clinically significant cardiovascular disease including but not limited to:

   * Unstable angina
   * Acute myocardial infarction within 6 months prior to screening
   * New York Heart Association (NYHA) Class II or greater congestive heart failure (see Section 20.6)
   * Clinically significant abnormalities in rhythm, conduction or morphology on resting ECG (e.g. complete left bundle branch block, third degree heart block)
   * Uncontrolled hypertension
   * Known LVEF < 50%
   * QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 msec for females and QTcF > 450 msec for males on screening electrocardiogram (ECG) or congenital long QT syndrome.
9. Participation in any other investigational trial at the time of informed consent signature.
10. Pregnant or lactating women.

    The following exclusion criteria applies to participants in Phase I:
11. Received anti-cancer therapy, including chemotherapy, immunotherapy, radiation therapy, biologic, herbal therapy, or any investigational therapy or investigational device, within 28 days (or 5 half-lives for biologic/non-cytotoxic agents, whichever is shorter), prior to the first dose of 177Lu-RAD204tr.
12. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-mediated AE.

    NOTE: endocrine immune-mediated AEs that are controlled with replacement therapy are allowed.
13. Has had or is scheduled to have major surgery < 28 days prior to the first dose of 177Lu-RAD204tr.Surgical procedures not considered to put participants at higher risk of AEs and/or interfere with the integrity of study outcome may be allowed on a case-by-case basis in discussion with the Sponsor.
14. Positive status for human immunodeficiency virus (HIV).
15. Active or chronic hepatitis B or C. Chronic hepatitis B or hepatitis C with undetectable viral loads on stable suppression therapy may be allowed on a case-by-case basis in discussion with study Sponsor.
16. Any medical condition which, in the opinion of the Investigator, places the participant at an unacceptably high risk for toxicities.
17. Any uncontrolled intercurrent illness or clinically significant uncontrolled condition(s), including but not limited to active bacterial, fungal, or viral infections requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time Activity Curves (TACs) | 72 hours
  Percent of the injected activity vs time for selected organs and tumors
Radiation dosimetry of Lu177-RAD204im | 72 hours
  Absorbed radiation doses of 177Lu-RAD204im in critical organs (e.g., kidneys, bone marrow)
Pharmacokinetics of 177Lu-RAD204im | 72 hours
  Half-life of 177Lu-RAD204im in blood
Biokinetics of 177Lu-RAD204im | 72 hours
  Time-integrated activity coefficients of 177Lu-RAD204im in organs and tumor lesions
Safety and tolerability of 177Lu-RAD204tr | 6 weeks
  The properties, incidence, nature and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Recommended dose(s) of 177Lu-RAD204tr for future exploration | 6 weeks
  Incidence of dose-limiting toxicities (DLTs) during the first 6 weeks following 177Lu-RAD204tr injection cycle of treatment

SECONDARY OUTCOMES:
Safety and tolerability of a single dose of 177Lu-RAD204im | 6 weeks
  The properties, incidence, nature and severity of AEs and SAEs per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Recommended dose(s) of 177Lu-RAD204im for future exploration | 2 weeks
  Incidence of dose-limiting toxicities (DLTs) in the first 2 weeks following 177Lu-RAD204im injection
Preliminary antitumor activity of 177Lu-RAD204tr | Up to 30 weeks
  Objective response rates (ORR) as assessed by RECIST v1.1
Radiation dosimetry of 177Lu-RAD204tr | 72 hours
  Absorbed radiation doses of 177Lu-RAD204tr in critical organs (e.g., kidneys, bone marrow)

OTHER OUTCOMES:
Level of agreement between 177Lu-RAD204im and standard of care imaging | Up to 30 weeks
  Standard of care imaging may include but is not limited to 18F-FDG-PET, CT-scan and/or 99mTc-MDP-bone
Effect of 177Lu-RAD204im and 177Lu-RAD204tr on tumor markers | Up to 30 weeks
  Circulating tumor DNA

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Cancer Research SA (CRSA), Adelaide, South Australia
  - GenesisCare Murdoch, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No